CLINICAL TRIAL: NCT06405139
Title: Phase II Study of Nanoliposomal Irinotecan, Oxaliplatin Plus Capecitabine As Conversion Therapy for Patients with Locally Advanced Colorectal Cancer
Brief Title: Nanoliposomal Irinotecan, Oxaliplatin Plus Capecitabine As Conversion Therapy of Locally Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4610
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: Locally Advanced Colorectal Cancer; Nanoliposomal Irinotecan; Oxaliplatin; Capecitabine; Conversion Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nanoliposomal Irinotecan, Oxaliplatin plus Capecitabine (Experimental): Patients will receive a modified FOLFOXIRI regimen (nanoliposomal irinotecan 60mg/m2, oxaliplatin 85 mg/m2, and capecitabine 800 mg/m2 twice daily, day 1 to 7), repeated every two weeks. The efficacy and resectability were evaluated every four cycles. Patients who had lesions that were radically resectable after evaluation will receive surgery. This medication will be administrated until disease progression or unacceptable toxicity or resectability or up to a maximum of 12 cycles.
  Interventions: Drug: Nanoliposomal Irinotecan, Oxaliplatin plus Capecitabine

INTERVENTIONS:
Drug: Nanoliposomal Irinotecan, Oxaliplatin plus Capecitabine — Nanoliposomal irinotecan 60mg/m2; Oxaliplatin 85 mg/m2; Capecitabine 800 mg/m2 twice daily, day 1 to 7; repeated every two weeks.
  Other Names: Nanoliposomal Irinotecan, Oxaliplatin, Capecitabine

SUMMARY:
Neoadjuvant chemotherapy has gained acceptance in treating locally advanced breast cancer, esophageal cancer, gastric cancer, and rectal cancer. However, the role of neoadjuvant chemotherapy for locally advanced colon cancer is still in the exploratory stage. The objective of this study is to explore the efficacy and safety of nanoliposomal irinotecan and oxaliplatin combined with capecitabine as a novel conversion therapy for locally advanced colorectal cancer patients.

DETAILED DESCRIPTION:
After patients are enrolled, they will receive a modified FOLFOXIRI regimen (nanoliposomal irinotecan 60mg/m2, oxaliplatin 85 mg/m2, and capecitabine 800 mg/m2 twice daily, day 1 to 7), repeated every two weeks. The efficacy and resectability were evaluated every four cycles. Patients who had lesions that were radically resectable after evaluation will receive surgery. This medication will be administrated until disease progression or unacceptable toxicity or resectability or up to a maximum of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. With a full understanding of the study, each participant volunteered to participate in this study and signed the informed consent (ICF) with good compliance and follow-up.
2. Age ≥18 and ≤70.
3. ECOG physical status score is 0 or 1.
4. Expected survival period ≥ 12 weeks.
5. Patients with histopathological confirmed MSS/pMMR-type adenocarcinoma of the colon and upper rectum which is not amenable to radiotherapy.
6. R0 resection was expected to be achieved by necessarily combined organ resection, or R0 resection cannot be achieved, assessed by CT and/or MRI and multidisciplinary team (MDT) discussion.
7. The clinical stage was cT4N1-2M0 or cT4bN0M0 according to AJCC 8th edition.
8. Patients with multiple primary colorectal cancer are eligible, if one of the primary tumors meets the inclusion criteria.
9. Patients with intestinal obstruction was relieved by colonic stenting or ostomy.
10. Patients had not received systematic therapy, such as surgery, chemotherapy, radiotherapy, targeted therapy, or immunotherapy.
11. At least one evaluable lesion (according to RECIST v1.1 standard);
12. Adequate organ function according to the following laboratory test values:

    1. Hemoglobin value ≥90g/L.
    2. White blood cell count ≥3.5*109/L.
    3. Absolute neutrophil count ≥1.5*109/L.
    4. Platelet count ≥100*109/L.
    5. Serum creatinine ≤ upper limit of normal (ULN) or creatinine clearance ≥60ml/min.
    6. Total serum bilirubin ≤1.5 upper normal limit (ULN).
    7. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5 upper limit of normal value (ULN).
13. Women with reproductive potential (< 2 years after the last menstrual period) and men use effective contraceptive methods until half a year after the last treatment.

Exclusion Criteria:

1. Patients who had shown hypersensitivity to the test drugs or other liposomal products.
2. Patients who have participated in other clinical trials in the past 4 weeks.
3. Previous or concurrent cancer diagnosed within 5 years (except cured basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix; the treatment of other malignant tumors has been completed for more than 5 years, and there is no clinical and imaging evidence of recurrence or progression except).
4. dMMR/MSI-H-type colorectal cancer.
5. Symptomatic peripheral neuropathy ≥ grade 2 (CTCAE 5.0).
6. Patients unable to swallow or lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
7. Patients had severe bleeding (CTCAE 5.0 grade ≥3) in the previous 4 weeks.
8. History of abdominal fistula, gastrointestinal perforation, intestinal obstruction, chronic diarrhea, or inflammatory bowel disease including Crohn's disease and ulcerative colitis within 6 months prior to the first study treatment.
9. Patients with interstitial lung disease, except only imaging demonstrated interstitial lung disease without symptoms.
10. Uncontrolled central nervous system metastasis (symptomatic or metastatic sites are midbrain, pons, medulla, or spinal cord) or other central nervous system diseases.
11. Received strong inhibitors or inducers of CYP3A4 and CYP2C8, or strong inhibitors of UGT1A1 in the previous 2 weeks.
12. Uncontrolled hypertension by a single-antihypertensive medication (systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg). Patients with severe cardiac dysfunction, such as LVEF< 50%, CHF≥ grade 2, severe/unstable angina, history of stroke or transient ischemic attack or myocardial infarction in the previous 6 months. Patients with a history of ventricular tachycardia, torsades de pointes, prolonged QTc, complete left bundle branch block, or third-degree atrioventricular conduction block.
13. Abnormal blood coagulation function, bleeding tendency or receiving thrombolysis or anticoagulant therapy.
14. Patients of childbearing potential are unwilling to practice contraception.
15. Patients with active hepatitis B, hepatitis C, syphilis, or human immunodeficiency virus infection.
16. Patients with current active infections require anti-infection treatment within 2 weeks of starting study treatment.
17. History of a definite neurological or mental disorder, including epilepsy and dementia.
18. Patients with any clinically significant disease, metabolic disorders, or laboratory abnormality. The investigator could reasonably consider those patients not suitable for the study, affecting the analysis of the results or putting those patients at high risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Organ-sparing R0 Resection Rate | 2 years
  The proportion of patients achieved R0 resection by only resecting the colon while other organs were retained.

SECONDARY OUTCOMES:
ypTNM stage | 2 years
  ypTNM stage evaluated by pathologists
TRG | 2 years
  Tumor regression grade evaluated by pathologists
R0, R1, R2 resection rate | 2 years
  R0, R1, R2 Resection Rate
Rate of residual or recurrent disease occurring within 2 years after surgery | 2 years
  The proportion of patients who experienced residual or recurrent disease within 2 years after surgery.
3-year OS rate | 3 years
  The proportion of patients achieved 3-year survival from treatment.
3-year PFS rate | 3 years
  The proportion of patients did not progress at least 3 years from treatment.
Safety and Tolerability | 2 years
  Incidence of Treatment-Related Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China